CLINICAL TRIAL: NCT04320745
Title: A Phase IV, Multi-center, Open-label, Single-arm 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Study of 16 Weeks Treatment With Androderm® in Hypogonadal Men
Brief Title: A Study to Evaluate Androderm®'s Effect on Blood Pressure in Adult Hypogonodal Male Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3146-402-016
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Androderm® 4 mg (Experimental): Participants received Androderm® 4 mg, transdermal dose, once daily (QD) for up to 16 weeks. At Day 14, if serum concentration was less than 400 nanograms per deciliter (ng/dL), the dose was increased to 6 mg, transdermal dose, QD for up to 16 weeks and if the serum concentration was more than 930 ng/dL, the dose was decreased to 2 mg, transdermal dose, QD for up to 16 weeks. The dose was not adjusted if serum concentrations were within the normal range.
  Interventions: Drug: Androderm®

INTERVENTIONS:
Drug: Androderm® — Androderm® transdermal dose.

SUMMARY:
This study will evaluate the effect of a once daily Androderm® dose on Blood Pressure (BP) in adult hypogonadal men as measured by 24-hour ABPM.

ELIGIBILITY:
Inclusion Criteria:

* Naïve to testosterone replacement, clomiphene, compounded or over-the-counter androgenic steroid derivatives, and dehydroepiandrosterone (DHEA), including investigational products that may affect the reproductive hormonal system or has not been treated with these compounds in the past 6 months
* Male participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period
* Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent
* Body mass index (BMI) < 35 kilograms per metre square (kg/m^2)
* Male

Exclusion Criteria:

* Uncontrolled systemic disease or clinically significant disease, in particular, liver, kidney or heart disease, including hypertension, congestive heart failure, coronary heart disease, chronic atrial fibrillation, sleep apnea or psychiatric illness, that in the investigator's opinion, would put the participant at an unacceptable risk with exposure to Androderm®
* History of prostate (current or in the past) or breast cancer
* Had a recent (within 2 years) history of stroke, transient ischemic attack, acute coronary event, venous thrombotic, or thromboembolic event
* History of alcohol or other substance abuse within the previous 2 years
* Known allergy or sensitivity to the study intervention or its components or other testosterone replacement medications
* Participant who works night shifts or who will need to perform strenuous manual labor while wearing the ABPM monitor

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 168 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (41):
- United States (41):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Coastal Clinical Research, LLC, An AMR Co., Mobile, Alabama
  - Urological Associates of South Arizona, PC, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Marvel Clinical Research, Huntington Beach, California
  - San Diego Clinical Trials, La Mesa, California
  - Wr-McCr, Llc, San Diego, California
  - Care Access Research, Santa Clarita, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Renstar Medical Research, Ocala, Florida
  - Ovieo Medical Research, LLC, Oviedo, Florida
  - Meridien Research, St. Petersburg, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Florida Urology Partners, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - Endocrine Consultants Newnan, Newnan, Georgia
  - Idoho Urologic Institute, Meridian, Idaho
  - The Iowa Clinic, West Des Moines, Iowa
  - DelRicht Research, LLC, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Bay State Clinical Trials, Inc, Watertown, Massachusetts
  - WR - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Premier Urology Group, Edison, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice, PLLC, New York, New York
  - Associated Urologist of North Carolina, Raleigh, North Carolina
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Academy of Diabetes Thyroid and Endocrine, El Paso, Texas
  - SMS Clinical Research, LLC2, Mesquite, Texas
  - AIM Trials, LLC, Plano, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Rainier Clinical Research Center, Inc, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Androderm® 4 mg
Started | 168
Completed | 121
Not Completed | 47
Not completed — Adverse Event | 26
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 12
Not completed — Protocol Deviation | 2
Not completed — Non-compliance With Study Drug | 2
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all treated participants who receive ≥ 1 administration of study intervention.
Groups:
- Androderm® 4 mg: Participants received Androderm® 4 mg, transdermal dose, QD for up to 16 weeks. At Day 14, if serum concentration was less than 400 ng/dL, the dose was increased to 6 mg, transdermal dose, QD for up to 16 weeks and if the serum concentration was more than 930 ng/dL, the dose was decreased to 2 mg, transdermal dose, QD for up to 16 weeks. The dose was not adjusted if serum concentrations were within the normal range.
Arm/Group | Androderm® 4 mg
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 136
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 28
  White | 133
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Average Systolic Blood Pressure (SBP) Obtained at Week 16
Description: SBP was collected by 24-hour ambulatory blood pressure monitoring (ABPM) device. 24-hour ABPM is defined as any assessment recorded at the specified analysis timepoint (baseline, Week 16) during the approximately 24-hour period after the ABPM device is applied through when the ABPM device is removed. BP parameters were collected at a minimum of 2 readings per hour for 24-hour recordings and were averaged.
Time Frame: Baseline and Week 16
Population: Modified Intent-to-treat (mITT) Population included all participants with valid baseline ABPM session of SBP, who received ≥ 1 administration of study intervention, ≥ 1 post-treatment assessments of SBP, valid Week 16 ABPM session of SBP, and at least 85% compliance to study intervention for the duration of the study.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Androderm® 4 mg
Number analyzed (Participants) | 62
millimeters of mercury (mmHg)
  Baseline | 123.2 (11.86)
  Change from Baseline at Week 16 | 3.5 (8.93)

2. Secondary Outcome: Change From Baseline in 24-hour Average Diastolic Blood Pressure (DBP) Obtained at Week 16
Description: DBP was collected by 24-hour ABPM device. 24-hour ABPM is defined as any assessment recorded at the specified analysis timepoint (baseline, Week 16) during the approximately 24-hour period after the ABPM device is applied through when the ABPM device is removed. BP parameters were collected at a minimum of 2 readings per hour for 24-hour recordings and were averaged.
Time Frame: Baseline and Week 16
Population: mITT Population included all participants with valid baseline ABPM session of SBP, who received ≥ 1 administration of study intervention, ≥ 1 post-treatment assessments of SBP, valid Week 16 ABPM session of SBP, and at least 85% compliance to study intervention for the duration of the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Androderm® 4 mg
Number analyzed (Participants) | 62
mmHg
  Baseline | 74.4 (7.16)
  Change from Baseline at Week 16 | 1.2 (5.43)

3. Secondary Outcome: Change From Baseline in 24-hour Average Mean Arterial Pressure (MAP) Obtained at Week 16
Description: MAP was collected by 24-hour ABPM device. 24-hour ABPM is defined as any assessment recorded at the specified analysis timepoint (baseline, Week 16) during the approximately 24-hour period after the ABPM device is applied through when the ABPM device is removed. BP parameters were collected at a minimum of 2 readings per hour for 24-hour recordings and were averaged.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Androderm® 4 mg
Number analyzed (Participants) | 62
mmHg
  Baseline | 90.4 (7.65)
  Change from Baseline at Week 16 | 1.7 (6.12)

4. Secondary Outcome: Change From Baseline in 24-hour Average Pulse Pressure Obtained at Week 16
Description: Pulse pressure was collected by 24-hour ABPM device. 24-hour ABPM is defined as any assessment recorded at the specified analysis timepoint (baseline, Week 16) during the approximately 24-hour period after the ABPM device is applied through when the ABPM device is removed. BP parameters were collected at a minimum of 2 readings per hour for 24-hour recordings and were averaged.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Androderm® 4 mg
Number analyzed (Participants) | 62
mmHg
  Baseline | 48.8 (8.90)
  Change From Baseline at Week 16 | 2.3 (4.82)

5. Secondary Outcome: Change From Baseline in 24-hour Average Heart Rate Obtained at Week 16
Description: Heart rate was collected by 24-hour ABPM device. 24-hour ABPM is defined as any assessment recorded at the specified analysis timepoint (baseline, Week 16) during the approximately 24-hour period after the ABPM device is applied through when the ABPM device is removed. BP parameters were collected at a minimum of 2 readings per hour for 24-hour recordings and were averaged.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Androderm® 4 mg
Number analyzed (Participants) | 62
beats per minute (bpm)
  Baseline | 72.4 (9.92)
  Change From Baseline at Week 16 | 2.2 (6.16)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of study or early termination visit (up to approximately 16 weeks)
Description: Safety Population included all treated participants who receive ≥ 1 administration of study intervention.
Arm/Group | Androderm® 4 mg
All-Cause Mortality (participants affected / at risk) | 0/168
Serious Adverse Events (participants affected / at risk) | 2/168
Other Adverse Events (participants affected / at risk) | 29/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androderm® 4 mg (N=168)
BRADYCARDIA (Cardiac disorders) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androderm® 4 mg (N=168)
APPLICATION SITE ERYTHEMA (General disorders) | 16 (26)
APPLICATION SITE RASH (General disorders) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04320745/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT04320745/SAP_001.pdf